CLINICAL TRIAL: NCT03904849
Title: A Pilot Human Laboratory Study of Cannabidiol in Alcohol Use Disorder
Brief Title: Cannabidiol for Alcohol Use Disorder
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was intended to produce pilot data for a center grant component that will no longer be conducted.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00086168
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (Active Comparator): Cannabidiol 6 mL of 100 mg/mL cannabidiol oral solution per day for 8 days
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Placebo 6 mL oral solution per day for 8 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol oral solution
  Other Names: Epidiolex
  Arms: Cannabidiol
Drug: Placebo — Placebo oral solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether cannabidiol, relative to placebo, affects subjective response to alcohol or alcohol drinking.

DETAILED DESCRIPTION:
This study will examine the effects of Epidiolex among adults who drink alcohol heavily but who are not seeking treatment for their alcohol use. Epidiolex is an FDA-approved formulation of cannabidiol, the primary non-psychoactive constituent of cannabis. Participants in the study will be randomly assigned to take Epidiolex or placebo for 8 days. There are 3 study visits, including a day-long visit in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for current Alcohol Use Disorder, as assessed by the Structured Clinical Interview for DSM-5 (SCID-5).
2. Reports drinking, on average, at least 20 standard alcoholic drinks per week for at least the past 3 months, with at least 5 standard alcoholic drinks during a drinking episode at least once per week during the past 3 months.
3. Currently not engaged in, and does not want treatment for, alcohol-related problems.
4. Age 21-40.
5. Able to read and understand questionnaires and informed consent.
6. Lives within 50 miles of the study site.

Exclusion Criteria:

1. Current DSM-5 diagnosis of any other substance use disorder except Nicotine Use Disorder.
2. Any psychoactive substance use (including cannabis, but excluding nicotine) within 30 days prior to screening, as indicated by self-report and urine drug screen.
3. Any cannabidiol use, in any formulation (e.g., oral, topical) within 30 days prior to screening.
4. Current DSM-5 Axis I diagnosis, including major depression, panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, bipolar affective disorder, schizophrenia, dissociative disorders, eating disorders, or any other psychotic or organic mental disorder.
5. Current active suicidal ideation, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS).
6. Current use of any psychoactive medication, any medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, topiramate), and/or antiepileptic medications (e.g., valproate).
7. Current use of any known hepatotoxic medication.
8. Current use of strong or moderate CYP3A4 inhibitors or inducers (commonly used examples not captured by other exclusion criteria include protease inhibitors, macrolide antibiotics [e.g., erythromycin], azole antifungals [e.g., ketoconazole], verapamil, and grapefruit juice).
9. Current use of strong or moderate CYP2C19 inhibitors or inducers (commonly used examples not captured by other exclusion criteria include proton pump inhibitors [e.g., omeprazole, lansoprazole], prednisone, and norethisterone).
10. History of severe alcohol withdrawal (e.g., seizure, delirium tremens), as evidenced by self-report and assessment with Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar).
11. Clinically significant medical problems such as cardiovascular, renal, gastrointestinal, or endocrine problems that would impair participation or limit medication ingestion.
12. Past alcohol-related medical illness, such as gastrointestinal bleeding, pancreatitis, or peptic ulcer.
13. Current or past hepatocellular disease, as indicated by: a) verbal report; b) Child-Pugh score > 6 (i.e., Child-Pugh class B or C); or c) alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin greater than the upper limit of the normal range at screening.
14. Females of childbearing potential who are pregnant (by serum HCG), nursing, or who are not using a reliable form of birth control.
15. Current charges pending for a violent crime (not including driving under the influence-related offenses).

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Average alcohol-induced sedation after medication ingestion | Average of measurements obtained 30, 60, 90, and 120 minutes following alcohol administration in the lab. Alcohol will be administered 2.5 hours after ingestion of study medication.
  Biphasic Alcohol Effects Scale sedation subscale score (range = 0-70; higher scores = greater sedation)
Average subjective response to alcohol after medication ingestion | Average of measurements obtained 30, 60, 90, and 120 minutes following alcohol administration in the lab. Alcohol will be administered 2.5 hours after ingestion of study medication.
  Subjective High Assessment Scale score (range = 0-130; higher scores = greater intoxication)

SECONDARY OUTCOMES:
Alcohol drinking in natural environment | 8 days of medication ingestion.
  Total number of standard drinks per day consumed during natural (usual environment) conditions

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Schacht, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No